CLINICAL TRIAL: NCT04950985
Title: A Multicentre Prospective Study to Improve Outcomes of Necrotising Otitis Externa in the UK
Brief Title: Improving Outcomes of Necrotising Otitis Externa
Acronym: IONOE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS:280342
Record Dates: First submitted 2021-06-25; First posted 2021-07-06 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Necrotising Otitis Externa
Keywords: infection; antimicrobials; otitis; externa
MeSH Terms: conditions — Infections; Otitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Selected sites will be asked to freeze any P. aeruginosa isolates routinely collected via ear swabs as part of clinical care from enrolled participants within 14 days of CT imaging. These de- identified samples may be sent from sites to undergo genotypic and phenotypic analysis at the University of Oxford for virulence factors to assess the relationship between these and disease severity. Of note, no samples beyond those routinely collected as part of the patients' care will be collected and no patient tissue samples will be stored. These samples will not contain any biological or genetic material from the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Adults undergoing a CT scan to investigate possible NOE.
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study — Observational study

SUMMARY:
A UK multi-centre prospective observational study of clinically possible cases of NOE.

DETAILED DESCRIPTION:
Patients with clinically possible NOE for whom CT imaging is requested will be recruited to the study by hospital staff at 20-25 UK sites.

NOE remains a relatively uncommon condition with UK - ENT surgeons report seeing between 1 and 10 cases per year. We plan to recruit 350 patients consented prior to or after CT imaging for a diagnosis of clinically possible NOE. After providing consent, patients will be asked to complete an EQ-5D-3L questionnaire. For patients consented remotely, this questionnaire will be completed via an interview. Local study staff will complete an online case report form hosted on Redcap™ for each patient including data on demographics, co-morbidities, clinical presentation, investigations and surgical and antibiotic management. Local study staff will review patients' hospital notes and contact patients' GPs by telephone 1-year post recruitment to assess clinical outcomes and mortality rates. Patients will then be contacted 12 months (+/- 1 month) post-recruitment by telephone by local study staff in order to confirm clinical outcomes (e.g. relapse) and gain information to complete the EQ-5D-3L questionnaire a second time.

All CT scans performed at recruitment and any other CT and/or MRI scans performed in the 12-month follow-up period will be de-identified and uploaded by local sites to an online, web-based secure repository for radiological images. Subspecialised radiologists blinded to clinical details will assess the images according to pre-agreed, standardised criteria.

Selected sites will be asked to freeze any P. aeruginosa isolates routinely collected via ear swabs as part of clinical care from enrolled participants within 14 days of CT imaging. These de-identified samples may be sent from sites to undergo genotypic and phenotypic analysis at the University of Oxford for virulence factors to assess the relationship between these and disease severity. Of note, no samples beyond those routinely collected as part of the patients' care will be collected and no patient tissue samples will be stored. These samples will not contain any biological or genetic material from the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old).
* Clinical diagnosis of possible NOE for whom CT imaging is requested or has been done as part of routine clinical care.

Exclusion Criteria:

* Any previous clinical diagnosis of NOE.
* CT performed or due to be performed at hospital other than recruiting study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be consented prior to or after CT imaging for a diagnosis of clinically possible NOE.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Demographic, management and outcome data | 12 months
  Describe the prevalence, demographics, clinical presentation, surgical and medical management and outcomes of clinically possible cases of NOE in the UK.

SECONDARY OUTCOMES:
Risk Factors for NOE | 12 months
  Identify risk factors for clinically possible NOE, SOE and definite NOE in the UK
Antibiotic Management of NOE | 12 months
  Understand whether differences in antibiotic choice and duration impact on clinical outcome of patients with SOE or NOE in the UK.
Role of Surgical Management in NOE | 12 months
  Describe the role of superficial sampling of the EAC, deep surgical sampling and debridement in cases of clinically possible NOE in the UK.
Economic Costs of NOE | 12 months
  Investigate the economic impact of clinically possible NOE in UK as measured by hospital bed days.
Affect of NOE on Generic Health Status | 12 months
  Assess changes in generic health status as measured using EQ-5D-3L in the year following enrolment of clinically possible NOE cases.
Radiological Changes of NOE | 12 months
  Assess agreement in interpretation of CT and/or MRI scans of clinically possible cases of NOE between locally reporting radiologists and blinded neuroradiology specialists working according to proposed standardised radiological criteria.
Pseudomonas Aeruginosa | 12 months
  Genotypic and phenotypic analysis of P. aeruginosa isolates to assess relationship between virulence markers and disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Hodgson, PhD, Principal Investigator — University of Oxford
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided